CLINICAL TRIAL: NCT01446289
Title: A Phase II Randomized, Observer-Blind, Multi-Center, Controlled Study of a Trivalent Group B Streptococcus Vaccine in Healthy Pregnant Women
Brief Title: Immune Response Induced by a Vaccine Against Group B Streptococcus and Safety in Pregnant Women and Their Offsprings
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V98_04; 2010-020840-36
Record Dates: First submitted 2011-09-27; First posted 2011-10-05 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Streptococcal Infection; Gram-positive Bacterial Infection; Bacterial Infection
Keywords: Group B streptococcus; GBS; Vaccine; Prevention of group B streptococcus infection
MeSH Terms: conditions — Streptococcal Infections; Gram-Positive Bacterial Infections; Bacterial Infections

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Group B Streptococcus Trivalent Vaccine (Experimental): Pregnant women who received one injection of Group B Streptococcus Trivalent Vaccine.
  Interventions: Biological: Group B Streptococcus Trivalent Vaccine
- Placebo (Placebo Comparator): Pregnant women who received one injection of saline solution.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Group B Streptococcus Trivalent Vaccine — Pregnant women who received one injection of Group B Streptococcus Trivalent Vaccine administered intramuscularly.
  Arms: Group B Streptococcus Trivalent Vaccine
Biological: Placebo — Pregnant women who received one injection of saline solution administered intramuscularly.
  Arms: Placebo

SUMMARY:
The study investigated the immune response induced by the Group B streptococcus vaccine in healthy pregnant women. In addition, the study investigated the amount of vaccine induced antibodies which were transferred to the newborn.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant women 18-40 years of age at 24-35 weeks of gestation at screening.
2. Individuals who have given a written consent after the nature of the study has been explained according to local regulatory requirements.
3. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.
4. Individuals who will be available for all scheduled visits (ie, not planning to leave the area before the end of the study period).

Exclusion Criteria:

1. Individuals who were unwilling and/or unable to give written informed consent to participate in the study.
2. Individuals with a history of severe allergic reactions after previous vaccinations such as anaphylactic shock, asthma, urticaria, or other allergic reaction or hypersensitivity to any vaccine component.
3. Individuals with any known or suspected impairment/alteration of immune function, either congenital or acquired or resulting from:

   * receipt of immunosuppressive therapy within 30 days prior to enrollment (any systemic corticosteroid administered for more than 5 days, or in a daily dose > 15 mg/kg/day prednisone or equivalent during any of 30 days prior to enrollment, or cancer chemotherapy).
   * receipt of immunostimulants.
   * receipt of parenteral immunoglobulin preparation, blood products, and /or plasma derivatives within 12 weeks prior to enrollment and for the full length of the study.

   Note: Anti-D (Rho) Immunoglobulins (anti-RhD) given for Anti-D prophylaxis were to be allowed.
4. Individuals characterized as "high risk" pregnancies at investigator discretion, such as those who have:

   * gestational diabetes
   * preeclampsia/eclampsia
   * women at risk of preterm labor (except positivity for vaginal GBS)
   * History of previous pregnancy complications including delivery of preterm infant.
   * History of still-birth, late abortions and children with congenital anomalies.
5. Individuals who had received any other investigational agent or investigational intervention during the course of the study.
6. Individuals with acute infection including oral temperature ≥ 38°C were to be temporarily excluded. They could be enrolled once the infection had resolved (as judged by investigator).
7. HIV positive by history.
8. Individuals reporting any known or suspected serious acute, chronic or progressive disease (eg, any history of neoplasm, malignancy, including lymphoproliferative disorder, diabetes, cardiac disease, malnutrition, renal failure, autoimmune disease, HBV or HCV, blood disorders).

   Note: Malignancies, highly likely to having been cured at the investigators discretion are allowed. (eg, no relapse since 5 years post last malignancy specific treatment).
9. Individuals with bleeding diathesis, or any condition that might have been associated with a prolonged bleeding time.
10. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, might have interfered with the subject's ability to participate in the study (eg, who were not able to comprehend or to follow all required study procedures for the whole period of the study).
11. Individuals with any progressive or severe neurologic disorder, seizure disorder, epilepsy or Guillain-Barré syndrome.
12. Individuals with history or any illness that, in the opinion of the investigator, might have posed additional risk to subjects due to participation in the study.
13. Individuals who were part of study personnel or close family members conducting this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines; Gilbert Donders, Prof., Principal Investigator — Regional Hospital Heilig Hart, Tienen, Belgium
Locations (5):
- Belgium (2):
  - UZ Leuven, Herestraat, Leuven
  - Regionaal Ziekenhuis Heilig Hart,, Gasthuismolenstraat 31, Tienen
- Canada (3):
  - University of British Columbia, Rm B3 25 B, 4500 Oak Street,, Vancouver, British Columbia
  - Dalhousie University, IWK Health Centre, 5850/5980 University Avenue,, Halifax, Nova Scotia
  - Centre hospitalier universitaire de Quebec (CHUQ)- hospital CHUL, Centre de recherche en infectiologie, 2705,, Boulevard Laurier, S-745, Quebec

REFERENCES:
- [Derived] Fabbrini M, Rigat F, Tuscano G, Chiarot E, Donders G, Devlieger R, Filippini S, Frigimelica E, Forte P, Wittke F, Halperin SA, Slobod K, Grandi G, Margarit I. Functional activity of maternal and cord antibodies elicited by an investigational group B Streptococcus trivalent glycoconjugate vaccine in pregnant women. J Infect. 2018 May;76(5):449-456. doi: 10.1016/j.jinf.2018.01.006. Epub 2018 Jan 31. PMID 29374589
- [Derived] Donders GG, Halperin SA, Devlieger R, Baker S, Forte P, Wittke F, Slobod KS, Dull PM. Maternal Immunization With an Investigational Trivalent Group B Streptococcal Vaccine: A Randomized Controlled Trial. Obstet Gynecol. 2016 Feb;127(2):213-21. doi: 10.1097/AOG.0000000000001190. PMID 26942345

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 centres.
Pre-assignment Details: A total of 86 pregnant subjects were enrolled in the study. 86 infants were enrolled in this study, delivered by 86 maternal subjects. There were 86 singleton deliveries.
Groups:
- Mothers GBS: Pregnant women who received one injection of GBS vaccine.
- Mothers Placebo: Pregnant women who received one injection of saline solution.
- Infants GBS: Infants born from mothers who received one injection of GBS vaccine.
- Infants Placebo: Infants born from mothers who received one injection of saline solution.
Period: Overall Study
Arm/Group | Mothers GBS | Mothers Placebo | Infants GBS | Infants Placebo
Started | 51 | 35 | 51 | 35
Completed | 50 | 35 | 50 | 35
Not Completed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled population
Groups:
- Total: Total of all reporting groups
Arm/Group | Mothers GBS | Mothers Placebo | Infants GBS | Infants Placebo | Total
Number analyzed (Participants) | 51 | 35 | 51 | 35 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] — Analysis was done on the enrolled population.
  years | 29.7 (4.9) | 30 (5.5) | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | 29.8 (5.1)
Age, Continuous [Mean (Standard Deviation); unit: days] — Analysis was done on the enrolled population.
  days | NA (NA) — presented elsewhere | NA (NA) — presented elsewhere | 0 (0) | 0 (0) | 0 (0)
Sex: Female, Male [Count of Participants; unit: Participants] — Analysis was done on the enrolled population.
  Participants
    Female | 51 | 35 | 21 | 15 | 122
    Male | 0 | 0 | 30 | 20 | 50
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 11 | 15 | 11 | 52
  Belgium | 36 | 24 | 36 | 24 | 120

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies in Mothers and Infants at Delivery/Birth
Description: GMCs of anti-Group B Streptococcus (GBS) capsular polysaccharide (CPS) antibodies against serotypes Ia, Ib and III in mothers and in infants at delivery/birth are presented.
Time Frame: Day of delivery/birth
Population: The analysis was done on the Immunogenicity Per Protocol Set (PPS), ie: all subjects in the enrolled population who correctly received the vaccine, provided evaluable serum samples at the relevant time points and had no major protocol violation as defined prior to un-blinding.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Mothers GBS | Mothers Placebo | Infants GBS | Infants Placebo
Number analyzed (Participants) | 45 | 30 | 45 | 30
µg/mL
  GBS Ia | 5.39 [2.97 to 9.77] | 0.41 [0.2 to 0.85] | 4.37 [2.39 to 7.99] | 0.4 [0.19 to 0.83]
  GBS Ib (N=40, 22, 40, 22) | 3.35 [1.44 to 7.77] | 0.064 [0.021 to 0.19] | 2.59 [1.14 to 5.87] | 0.092 [0.032 to 0.27]
  GBS III (N=40, 25, 40, 25) | 2.45 [1.15 to 5.2] | 0.056 [0.022 to 0.14] | 1.65 [0.78 to 3.5] | 0.055 [0.022 to 0.14]

2. Primary Outcome: Geometric Mean of the Ratios Between Infant Antibody Level (μg/mL) and Maternal Antibody Level (μg/mL) at Time of Delivery
Description: The Geometric mean transfer ratio of anti-GBS CPS antibodies against serotypes Ia, Ib and III at delivery is calculated as the geometric mean of the pairwise ratios between the antibody concentrations from infant at birth and to maternal serum concentration at delivery.
Time Frame: Day of delivery/birth
Population: The analysis was done on the Immunogenicity PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Mothers GBS | Mothers Placebo
Number analyzed (Participants) | 45 | 30
Ratio
  GBS Ia | 0.81 [0.72 to 0.91] | 0.97 [0.85 to 1.11]
  GBS Ib (N=40, 22) | 0.77 [0.62 to 0.97] | 1.44 [1.06 to 1.94]
  GBS III (N=40, 25) | 0.68 [0.59 to 0.78] | 0.99 [0.83 to 1.18]

3. Secondary Outcome: GMCs (Enzyme-linked Immunosorbent Assay, ELISA) Antibodies Against Serotypes Ia, Ib and III in Maternal Subjects
Description: GMCs (ELISA) of anti-GBS CPS antibodies against serotypes Ia, Ib and III in maternal subjects at study day 1, study day 31 and at day 91 post-partum after one administration of GBS vaccine or placebo are reported.
Time Frame: Day 1, day 31 and day 91 post-delivery
Population: The analysis was done on the Immunogenicity PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Mothers GBS | Mothers Placebo
Number analyzed (Participants) | 51 | 35
µg/mL
  GBS Ia (day 1) | 0.28 [0.19 to 0.41] | 0.37 [0.24 to 0.58]
  GBS Ia (day 31; N=49, 32) | 4.83 [2.89 to 8.06] | 0.36 [0.19 to 0.65]
  GBS Ia (day 91 post-delivery; N = 44, 34) | 5.89 [3.86 to 8.99] | 0.46 [0.29 to 0.75]
  GBS Ib (day 1; N= 50, 34) | 0.13 [0.084 to 0.19] | 0.084 [0.051 to 0.14]
  GBS Ib (day 31; N=49, 31) | 1.68 [0.97 to 2.92] | 0.14 [0.069 to 0.27]
  GBS Ib (day 91 post-delivery; N= 44, 33) | 3.46 [2.33 to 5.14] | 0.17 [0.11 to 0.27]
  GBS III (day 1) | 0.11 [0.07 to 0.16] | 0.093 [0.056 to 0.15]
  GBS III (day 31; N= 49, 32) | 1.46 [0.83 to 2.57] | 0.12 [0.06 to 0.23]
  GBS III (day 91 post-delivery; N=44, 34) | 2.69 [1.78 to 4.06] | 0.11 [0.07 to 0.18]

4. Secondary Outcome: Geometric Mean Ratios (GMRs) of Antibody GMCs (ELISA) in Maternal Subjects
Description: GMRs of GMCs (ELISA) of anti-GBS CPS antibodies against serotypes Ia, Ib and III, in maternal subjects at study day 31, at delivery and at day 91 post-partum versus day 1 (baseline) after one administration of GBS vaccine or placebo are reported.
Time Frame: Day 31, day of delivery, day 91 post-delivery
Population: The analysis was done on the Immunogenicity PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Units Other Than Participants: strains
Arm/Group | Mothers GBS | Mothers Placebo
Number analyzed (Participants) | 51 | 35
Number analyzed (strains) | 110 | 110
Ratio
  GBS Ia (Day 31/day 1; N=49, 32) | 15 [9.12 to 25] | 1.22 [0.66 to 2.25]
  GBS Ia (Delivery/day 1) | 16 [11 to 25] | 1.2 [0.72 to 2.01]
  GBS Ia (day 91 post-delivery/day 1; N= 44, 34) | 19 [12 to 28] | 1.51 [0.94 to 2.42]
  GBS Ib (Day 31/day 1; N=48, 30) | 18 [9.94 to 32] | 1.14 [0.56 to 2.35]
  GBS Ib (Delivery/day 1; N=50, 34) | 23 [14 to 39] | 1.13 [0.63 to 2.05]
  GBS Ib (day 91 post-delivery/day 1; N=44, 32) | 33 [22 to 48] | 1.53 [0.96 to 2.43]
  GBS III (Day 31/day 1; N=49, 32) | 17 [9.17 to 30] | 1.19 [0.59 to 2.42]
  GBS III (Delivery/day 1) | 20 [12 to 33] | 1.08 [0.6 to 1.96]
  GBS III (day 91 post-delivery/day 1; N=44, 34) | 28 [18 to 43] | 1.11 [0.69 to 1.8]

5. Secondary Outcome: GMC (ELISA) of Anti-GBS CPS Antibodies in Infants
Description: GMC (ELISA) of anti-GBS CPS antibodies against serotypes Ia, Ib and III in infants at birth and at 3 months of age are reported.
Time Frame: Day of birth and day 91 after birth
Population: The analysis was done on the Immunogenicity PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Infants GBS | Infants Placebo
Number analyzed (Participants) | 35 | 25
μg/mL
  GBS Ia (day of birth) | 5.14 [2.64 to 10] | 0.33 [0.15 to 0.71]
  GBS Ia (day 91 after birth) | 1.28 [0.76 to 2.16] | 0.25 [0.13 to 0.46]
  GBS Ib (day of birth; N=31, 20) | 2.93 [1.14 to 7.57] | 0.1 [0.031 to 0.32]
  GBS Ib (day 91 after birth) | 0.54 [0.25 to 1.19] | 0.063 [0.025 to 0.16]
  GBS III (day of birth; N=30, 22) | 1.93 [0.82 to 4.59] | 0.065 [0.024 to 0.18]
  GBS III (day 91 after birth) | 0.43 [0.21 to 0.86] | 0.065 [0.029 to 0.15]

6. Secondary Outcome: GMRs of Anti-GBS CPS Antibody GMCs (ELISA) in Infants at 3 Months of Age Versus GMCs at Birth
Description: GMRs of anti-GBS CPS antibody GMCs (ELISA) against serotypes Ia, Ib and III in infants at 3 months of age (day 91 after birth) versus GMCs at birth are reported.
Time Frame: Day 91 after birth
Population: The analysis was done on the Immunogenicity PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Infants GBS | Infants Placebo
Number analyzed (Participants) | 35 | 25
Ratio
  GBS Ia | 0.25 [0.19 to 0.32] | 0.76 [0.57 to 1.01]
  GBS Ib (N=31, 20 ) | 0.22 [0.16 to 0.29] | 0.54 [0.38 to 0.78]
  GBS III (N=30, 22) | 0.25 [0.19 to 0.32] | 0.85 [0.62 to 1.16]

7. Secondary Outcome: Percentages of Infant Subjects Showing Anti-diphtheria Antibodies GMCs (ELISA) Over 0.1 IU/mL at 1 Month After the Last Routine Infant Immunization
Description: Percentages of infant subjects showing anti-diphtheria antibodies GMCs (ELISA) over 0.1 IU/mL in sera collected at 1 month after the last routine infant immunization (ie, either 5 months or 7 months after birth, depending on the vaccination schedule) are reported.
Time Frame: 1 month after the last routine infant immunization
Population: The analysis was done on the Immunogenicity PPS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Infants GBS | Infants Placebo
Number analyzed (Participants) | 40 | 27
Percentages of subjects | 100 [91 to 100] | 100 [87 to 100]

8. Secondary Outcome: Percentage of Maternal Subjects Reporting Solicited Local and Systemic Adverse Events (AEs)
Description: Percentage of maternal subjects reporting solicited local and systemic AEs and other indicators of reactogenicity from day 1 to 7 after vaccination are reported.
Time Frame: From day 1 to 7 after vaccination
Population: The analysis was done on the Safety Set, ie, all subjects in the enrolled population who received a study vaccination, provided post vaccination safety data, provided post-baseline safety data.
Measure: Number; unit: Percentages of subjects
Arm/Group | Mothers GBS | Mothers Placebo
Number analyzed (Participants) | 50 | 34
Percentages of subjects
  Any local | 40 | 24
  Induration (>=25 mm; N =49, 34) | 6 | 0
  Swelling (>=25 mm; N =49, 34) | 4 | 0
  Ecchymosis (>=25 mm; N =49, 34 ) | 2 | 0
  Erythema (>=25 mm; N =49, 34) | 6 | 0
  Pain (N =49, 34) | 35 | 12
  Any systemic | 46 | 38
  Chills (N =49, 34) | 4 | 3
  Fatigue (N =49, 34) | 31 | 26
  Malaise (N =49, 34) | 14 | 9
  Myalgia (N =49, 34) | 27 | 3
  Headache (N =49, 34) | 16 | 21
  Rash (N =49, 34) | 2 | 3
  Arthralgia (N =49, 34) | 4 | 9
  Nausea (N =49, 34) | 6 | 9
  Fever, body temperature >38° C (N =49, 33) | 0 | 0
  Any other | 8 | 3
  Stayed home (N =49, 34) | 2 | 0
  Use of analgesics/antipyretics (N =49, 34) | 6 | 3

9. Secondary Outcome: Percentage of Maternal Subjects Reporting Unsolicited AEs and Serious Adverse Events (SAEs)
Description: Percentage of maternal subjects reporting unsolicited AEs, SAEs, AEs requiring a non-routine physician's visit, AEs leading to withdrawal are reported.
Time Frame: All AEs were recorded until delivery, after delivery all AEs requiring a non-routine physician's visit and AEs leading to withdrawal from the study. SAEs were collected for the duration of the trial.
Population: The analysis was done on the Safety Set.
Measure: Number; unit: Percentages of subjects
Arm/Group | Mothers GBS | Mothers Placebo
Number analyzed (Participants) | 51 | 35
Percentages of subjects
  Any unsolicited AE | 63 | 74
  Any SAE | 14 | 23
  Medically-attended AEs | 51 | 54
  AEs leading to withdrawal | 0 | 0

10. Secondary Outcome: Percentages of Infants Reporting SAEs
Description: Percentages of infants born from women who received either one injection of the study vaccine or placebo, reporting SAEs from birth until study termination are reported.
Time Frame: From birth until study termination
Population: The analysis was done on the Safety Set.
Measure: Number; unit: Percentages of subjects
Arm/Group | Infants GBS | Infants Placebo
Number analyzed (Participants) | 51 | 35
Percentages of subjects | 24 | 31

ADVERSE EVENTS:
Time Frame: Solicited (systematic) AEs were collected from day 1 to 7 after vaccination; unsolicited (non-systematic) AEs from day 1 until delivery, SAE from day 1 until study termination (day 151 for subjects enrolled in Belgium, day 211 for subjects in Canada).
Description: The analysis was done on the Safety Set.
Groups:
- Mothers GBS: Pregnant women who received one dose of GBS vaccine.
- Infants GBS: Infants born from mothers who received one dose of GBS vaccine.
Arm/Group | Mothers GBS | Mothers Placebo | Infants GBS | Infants Placebo
Serious Adverse Events (participants affected / at risk) | 7/51 | 8/35 | 12/51 | 11/35
Other Adverse Events (participants affected / at risk) | 35/51 | 24/35 | 0/51 | 2/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mothers GBS (N=51) | Mothers Placebo (N=35) | Infants GBS (N=51) | Infants Placebo (N=35)
Renal hypoplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Jaundice acholuric (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cataract congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Renal dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Crying (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 1
Sepsis neonatal (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 1
Post procedural haemorrage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foetal monitoring (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Unstable foetal lie (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0
Postpartum depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal hypertrophy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cervix disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal haemorrage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tachipnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Caesarean section (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mothers GBS (N=51) | Mothers Placebo (N=35) | Infants GBS (N=51) | Infants Placebo (N=35)
Haemorrhoids (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 0 | 0
Fatigue (General disorders) | 15 | 10 | 0 | 0
Injection site erythema (General disorders) | 9 | 4 | 0 | 0
Injection site haemorrhage (General disorders) | 2 | 3 | 0 | 0
Injection site induration (General disorders) | 6 | 1 | 0 | 0
Injection site pain (General disorders) | 18 | 8 | 0 | 0
Injection site swelling (General disorders) | 4 | 1 | 0 | 0
Malaise (General disorders) | 7 | 4 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 0 | 0
Cystitis (Infections and infestations) | 2 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 10 | 0 | 0
Postpartum depression (Psychiatric disorders) | 1 | 2 | 0 | 0
Vaginal haemorrage (Reproductive system and breast disorders) | 1 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.